CLINICAL TRIAL: NCT02122328
Title: USFetus Randomized Clinical Trial: Sequential vs. Standard Laser Treatment of Twin-twin Transfusion Syndrome
Brief Title: Sequential vs. Standard Laser Treatment of Twin-twin Transfusion Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Ramen Chmait, Associate Professor, Clinical Obstetrics & Gynecology, Pediatrics, and Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-09-00680
Record Dates: First submitted 2014-04-16; First posted 2014-04-24 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Twin Twin Transfusion Syndrome
Keywords: Twin twin transfusion syndrome; Sequential laser photocoagulation of communicating vessels
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selective procedure (Active Comparator): Selective laser photocoagulation of communicating vessels.
  Interventions: Procedure: Selective laser photocoagulation of communicating vessels
- Sequential procedure (Experimental): Sequential laser photocoagulation of communicating vessels
  Interventions: Procedure: Sequential laser photocoagulation of communicating vessels.

INTERVENTIONS:
Procedure: Sequential laser photocoagulation of communicating vessels.
  Arms: Sequential procedure
Procedure: Selective laser photocoagulation of communicating vessels
  Arms: Selective procedure

SUMMARY:
The investigators hypothesize that treatment of twin-twin transfusion syndrome (TTTS) using sequential laser photocoagulation of communicating vessels (SQLPCV) over the predominant method, selective laser photocoagulation of communicating vessels (SLPCV), may provide vascular stability to the donor fetus. The primary objective is to evaluate the perinatal outcome, specifically, donor intrauterine survival of TTTS managed by SQLPCV vs. SLPCV in a prospective, randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age: 16 weeks, 0 days to 26 weeks, 0 days.
* Confirmed TTTS patients, who by definition meet the following sonographic criteria:

  * Single placenta.
  * Polyhydramnios: maximum vertical pocket ≥ 8 cm in the recipient twin, prior to amniodrainage.
  * Oligohydramnios: maximum vertical pocket ≤ 2 cm in the donor twin, prior to amniodrainage.
  * Thin dividing membrane (absence of twin peak sign) or absence of dividing membrane (monoamniotic).
  * Same gender, if visible.
  * Quintero Stages 1-4.
* Patients choosing laser therapy that have undergone prior therapeutic amniocentesis may be included.
* Patients with an anterior placenta may be included.
* Triplet gestations with two or three fetuses sharing the same placenta may be included.
* Patients must be able to give written informed consent.

Exclusion Criteria:

* Patients unable or unwilling to participate in the study or to be followed up.
* Patients unable to give written informed consent.
* Presence of major congenital anomalies that may not warrant surgery.
* Known unbalanced chromosomal complement.
* Prior intentional septostomy (purposely making a hole in the dividing membrane).
* Ruptured membranes.
* Chorioamnionitis.
* Abnormal intracranial ultrasound findings of either fetus to include, but not limited to: intraventricular hemorrhage, porencephalic cysts, hydrocephalus, Dandy-Walker syndrome, holoprosencephaly and agenesis of the corpus callosum. Isolated ventriculomegaly (atrium 10-19 mm) may or may not be used as exclusion criteria.
* Placental abruption.
* Active labor.
* Patient unwilling to receive blood products.
* Recipient twin with a middle cerebral artery peak systolic velocity > 1.5 multiples of the median (indicative of fetal anemia).
* Any other patient deemed inappropriate for the study by the principal investigator.

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 642 (Actual)
Dates: Start 2010-06-09 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
To compare donor intrauterine survival (alive at birth) for those undergoing SQLPCV vs. SLPCV. | Birth
  A comparison of donor survival at birth will be made between subjects assigned to the sequential (SQLPCV) procedure versus those assigned to the selective (SLPCV) procedure.

SECONDARY OUTCOMES:
Surgical complications | 21 post-operative days

OTHER OUTCOMES:
Fetal/neonatal/infant outcomes | Birth to 6 months of life

CONTACTS AND LOCATIONS:
Overall Officials: Ramen Chmait, MD, Principal Investigator — University of Southern California
Locations (1):
- Hollywood Presbyterian Medical Center, Los Angeles, California, United States